CLINICAL TRIAL: NCT01828424
Title: Prediction of Postoperative Pain by Measuring Nociception at the End of Surgery
Acronym: PREPOP
Status: Completed | Type: Observational
Sponsor: Benno Rehberg-Klug (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor-Investigator, Benno Rehberg-Klug, médecin adjoint agrégé, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: CER 12-262
Record Dates: First submitted 2013-04-03; First posted 2013-04-10 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Acute Postoperative Pain
Keywords: acute pain
MeSH Terms: conditions — Pain, Postoperative; Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There is a large variability of postoperative pain intensity and of the drug doses necessary to alleviate this pain. The investigators hypothesis is that a measurement of nociception at the end of surgery, using either the RIII reflex threshold, measures of heart rate variability or the pupil dilatation reflex measured by pupillometry, in relation to the doses of opioids used intraoperatively will yield a prediction of postoperative pain.

DETAILED DESCRIPTION:
Acute postoperative pain needs to be alleviated quickly to avoid sensitization in the postoperative period, since sensitization can lead to pain chronification. Severe acute postoperative pain is the most important risk factor in the development of persistent postoperative pain.

Unfortunately, the dose of opioids necessary to alleviate postoperative pain is highly variable, even between patients having been exposed to the same surgical procedure. Anesthesiologists usually try to prevent immediate postoperative pain by adjusting analgesic dosing at the end of surgery to the perceived need of analgesia. However, this approach is limited by the problem of respiratory depression induced by a too large dose of opiate analgesics. Studies have shown that despite these attempts many patients awake with moderate to severe pain.

A means of predicting immediate postoperative pain after surgery and the response to opiate analgesics would therefore be highly desirable. Many studies have tried to reveal predictive factors which can be evaluated before the start of the surgery, but these can explain only about 50% of the observed variability in postoperative pain intensity.

A different approach may be the evaluation of intraoperative nociception at the end of surgery to directly guide appropriate analgesia before the patient has regained consciousness. Measuring reflex pupil dilation after a standardized electrical stimulus is one method to measure opioid effect intra-operatively. This parameter may reflect opioid sensitivity, but not pain sensitivity.

The primary objective of this study is the evaluation of measures of nociception such as the pupillary dilation reflex or heart rate variability on acute pain after surgery.

In addition, pupillary dilation reflex and heart rate variability will be evaluated in their predictive performance of blood pressure and heart rate changes due to intubation.

The study is designed as a single centre, observational, descriptive study.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) physical status less than 3
* Able to read and understand the information sheet and to sign and date the consent form
* Being scheduled for elective gynaecological intraperitoneal surgery (laparoscopy, laparoscopic hysterectomy, vaginal hysterectomy, abdominal hysterectomy) under general anesthesia
* Age>18

Exclusion Criteria:

* Regional anesthesia (epidural analgesia, multi-orifice wound catheter, or transversus abdominis plane block) used for postoperative analgesia
* Surgery performed under regional anesthesia
* Contraindication to a general anesthesia using propofol and sufentanil (e.g. necessity for rapid sequence induction)
* BMI >35 (limit of the equations used in the target controlled infusion device)
* Severe renal insufficiency precluding use of morphine (GFR<30 ml/min)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for elective gynaecological intraperitoneal surgery (laparascopy, laparoscopic hysterectomy, vaginal hysterectomy, abdominal hysterectomy) under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
pain upon arrival in the recovery room | 20 minutes
  presence or absence of pain reported by the patient upon arrival in the recovery room
opioid effect | 20 minutes
  Opioid effect as defined on a scale of -1 to +1:
  "+1" =pain intensity >3 upon arrival in the recovery room, necessitating treatment "0" = pain intensity <=3 upon arrival in the recovery, no respiratory depression at the time of stop of the sufentanil infusion (respiratory frequency immediately >8/min) "-1" = pain intensity <=3 upon arrival in the recovery, time to a steady respiratory frequency of >8/min is less than 20 min (=mean of all patients) from time of stop of the sufentanil infusion. This outcome will be used as primary outcome if less than 20% of patients report a pain intensity of >3 upon arrival in the recovery room.

SECONDARY OUTCOMES:
respiratory depression | 20 minutes
  The time from the stop of the sufentanil infusion until a steady respiratory rate of >8/min has been reached
cumulative morphine dose | 24 hours
  The cumulative morphine at 2h, 12h and at 24h after the end of surgery (intravenous nurse administered doses in the recovery room and consumption measured by the patient-controlled analgesia pump)
systolic blood pressure increase after intubation | 6 minutes
  change in systolic blood pressure during the 3 minutes following intubation compared to the 3 minutes before intubation
heart rate increase after intubation | 6 minutes
  change in heart rate during the 3 minutes following intubation compared to the 3 minutes before intubation
mean pain intensity first 24h | 24h
  mean of the 3 pain intensity measurements on the ward during the first 24 postoperative hours, after discharge from the recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Benno Rehberg-Klug, MD, Study Director — Department of anesthesiology, HUG
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

REFERENCES:
- [Background] von Dincklage F, Hackbarth M, Mager R, Rehberg B, Baars JH. Monitoring of the responsiveness to noxious stimuli during anaesthesia with propofol and remifentanil by using RIII reflex threshold and bispectral index. Br J Anaesth. 2010 Feb;104(2):201-8. doi: 10.1093/bja/aep357. Epub 2009 Dec 22. PMID 20031950